CLINICAL TRIAL: NCT05820100
Title: A Prospective Multi-Center Observational Study to Assess the Reliability and Validity of the Multi-Luminance Y-Mobility Test (MLYMT) and Multi-Luminance Shape Discrimination Test (MLSDT)
Brief Title: Observational Study to Assess the Reliability and Validity of the MLYMT and MLSDT
Status: Completed | Type: Observational
Sponsor: Nanoscope Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NTXOBS-001
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Retinitis Pigmentosa; Retinal Dystrophy
Keywords: Retinitis Pigmentosa; Inherited Retinal Diseases; Eye Diseases; Retinal Degeneration; Mobility Test; Multi-luminance Y- Mobility Test
MeSH Terms: conditions — Retinitis Pigmentosa; Retinal Dystrophies; Eye Diseases; Retinal Degeneration | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normally Sighted: Participants with clinically normal ocular findings and BCVA better than logMAR 0.3 in each eye.
  Interventions: Other: Observational
- Severely Sight Impaired: Participants with BCVA no better than logMAR 1.6 in better seeing eye, and worse than logMAR 1.9 in the worse seeing eye, and a clinical diagnosis of advanced RP
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — The goal of this observational study is to assess the reliability and validity of the multi-luminance Y-Mobility Test (MLYMT) and multi-luminance shape description test (MLSDT) for evaluation of subjects with severe vision impairment due to RP.
  Normally sighted subjects will provide a control group. The MLYMT consists of two LED panels, one of which is illuminated at multiple luminance levels, positioned at the end of Y-configuration. Seven obstacles are placed ahead of the panels, which the test subject should detect and avoid before reaching and touching the lit panel.

SUMMARY:
This is a prospective Multi-Center Observational Study to assess the reliability and validity of the Multi-Luminance Y-Mobility Test (MLYMT) and Multi-Luminance Shape Discrimination Study (MLSDT) Main Outcome Measures: (i) Performance scores in normal and severely visually impaired subjects with a clinical diagnosis of retinitis pigmentosa (RP) on MLYMT and MLSDT at multiple luminance levels and (ii) reliability and content validity of MLYMT and MLSDT.

DETAILED DESCRIPTION:
Two assessment visits will be conducted in order to evaluate functional visual performance in severely vision impaired subjects with RP and normally sighted subjects. Two visits will occur at week 0 and week 4 with functional vision assessments occurring at both visits in order to assess visit-to-visit variability. For the MLYMT, navigational vision will be assessed using each eye and binocularly at up to 6 different light levels (range 0.3 to 100 lux). Subjects will also perform the Multi-Luminance Shape Discrimination Test (MLSDT) which assesses near object recognition under different lighting levels. MLYMT and MLSDT performance will be evaluated together with Best Corrected Visual Acuity (BCVA), Visual Field (VF) and responses to visual function questionnaires. Subjects will be assigned to one of two cohorts based on presence or absence of RP in addition to BCVA performance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Able to comprehend and give informed consent.
3. Able to comply with testing and all protocol tests.
4. Eligible for 1 of 2 cohorts listed below:

Cohort 1: Normally Sighted Participants with clinically normal ocular findings and BCVA better than logMAR 0.3 (as confirmed by ETDRS letter score > 73) in each eye Cohort 2: Severely Sight Impaired Participants with BCVA no better than logMAR 1.6 in better seeing eye, and worse than LogMAR 1.9 in the worse seeing eye, and a clinical diagnosis of advanced RP

Exclusion Criteria:

1. Concurrent participation in any interventional clinical trial or receipt of an investigational drug within the previous 6 months
2. Presence of any condition other than RP Disease that impairs visual acuity or visual fields e.g., visually significant cataract or visual field loss in glaucoma
3. Presence of neurological condition that impairs visual acuity or visual field, e.g., hemianopia secondary to stroke
4. Individuals who refuse or are incapable of performing mobility testing
5. Individuals with retinal prosthesis (such as ARGUS-II)
6. Participation in Nanoscope studies NTXMCO-002 (RESTORE) or NTXMCO-004 (STARLIGHT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 35 adult subjects, to one of 2 cohorts. Subjects who meet all the inclusion criteria and for whom none of the exclusion criteria apply will be eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-10-17 (Actual)

PRIMARY OUTCOMES:
MLYMT scores in normal and severely visually impaired subjects with a clinical diagnosis of RP on MLYMT | 4 Weeks
  A higher MLYMT score (range -1 to 5) indicates better navigational vision.
MLSDT scores in normal and severely visually impaired subjects with a clinical diagnosis of RP on MLSDT | 4 Weeks
  A higher MLSDT score (range 0 to 5) indicates greater shape discrimination ability at lower luminance level
Reliability and construct validity of MLYMT | 4 Weeks
  Evaluation of the performance (test-retest reliability) of the test(s) based on the visual acuity
Reliability and construct validity of MLSDT | 4 Weeks
  Evaluation of the performance (test-retest reliability) of the test(s) based on the visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Dr Samarendra Mohanty, Study Chair — Nanoscope Therapeutics Inc.
Locations (8):
- United States (7):
  - Nanoscope Clinical Site, Phoenix, Arizona
  - Nanoscope Clinical Site, Beverly Hills, California
  - Nanoscope Clinical Site, Miami, Florida
  - Nanoscope Clinical Site, Fargo, North Dakota
  - Nanoscope Clinical Site, Bellaire, Texas
  - Nanoscope Clinical Site, McAllen, Texas
  - Nanoscope Clincal Site, San Antonio, Texas
- Nanoscope Clinical Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
The results of the clinical trial will be made available when the study is completed. The results will be published on this site and be available to conference presentations and publications.
Time Frame: 12 months after the study is completed
Access Criteria: Reliability and Validity of MLYMT and MLSDT